CLINICAL TRIAL: NCT07081776
Title: Evaluation of the Effects on Carbon Dioxide (paCO2) of a New Oronasal Mask in Patients With Severe Exacerbation of COPD Requiring Non-Invasive Mechanical Ventilation: A Single-Center, Exploratory, Randomized Cross-Over Study
Brief Title: Evaluation of the Effects on Carbon Dioxide (paCO2) of a New Oronasal Mask in Patients With Severe COPD Exacerbation Requiring Non-Invasive Mechanical Ventilation
Acronym: OPTIMUS-MASK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Bologna (Other); Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, dr. Stefano Nava, Prof., IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMUS-MASK
Record Dates: First submitted 2025-04-28; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: COPD; Respiratory Acidosis
Keywords: COPD; NIV; Oronasal Mask; PaCO2
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Acidosis, Respiratory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OptiNIV (Experimental): Patients will undergo treatment with the OptiNIV Mask
  Interventions: Device: OptiNIV
- Visairo (Active Comparator): Patients will undergo treatment with Visairo Mask
  Interventions: Device: Visairo

INTERVENTIONS:
Device: OptiNIV — Patients assigned to the "OptiNIV" group will be submitted to two consecutive 60-minute sessions. In the first session, they will receive NIV with an "optimized" mask (OptiNIV) and in the second session they will receive NIV with a traditional" oronasal mask (Visairo). The study will follow a crossover design, meaning each patient will undergo both sessions, In both sessions, NIV will be delivered using the same ventilator (ASTRAL 150 - ResMed Europe). Ventilator settings will be set to ensure the most effective ventilation and the best comfort for each patient. However, these settings must remain unchanged during the two sessions. A 30-minute washout period is planned between the sessions, during which patients will receive traditional oxygen therapy through a Venturi mask. The 30 min wash-out periodod can be extended until PtCO₂ returns within ±2 mmHg of baseline or until 60 minutes have passed. The maximum total treatment time for each patient will be approximately 3 hours.
  Arms: OptiNIV
Device: Visairo — Patients assigned to the "Visairo" group will be submitted to two consecutive 60-minute sessions. In the first session, they will receive NIV with a "traditional" oronasal mask (Visairo) and in the second session they will receive NIV with an "optimized" mask (OptiNIV). The study will follow a crossover design, meaning each patient will undergo both sessions. In both sessions, NIV will be delivered using the same ventilator (ASTRAL 150 - ResMed Europe). Ventilator settings will be set to ensure the most effective ventilation and the best comfort for each patient. However, these settings must remain unchanged during the two sessions. A 30-minute washout period is planned between the sessions, during which patients will receive traditional oxygen therapy through a Venturi mask. The 30 min wash-out periodod can be extended until PtCO₂ returns within ±2 mmHg of baseline or until 60 minutes have passed. The maximum total treatment time for each patient will be approximately 3 hours.
  Arms: Visairo

SUMMARY:
This single-center, crossover study aims to investigate the effects of the new OptiNIV oronasal mask used during NIV in COPD patients with respiratory acidosis following an exacerbation. The goal is to evaluate whether the clinical benefits, in terms of reducing PaCO2 levels, are greater with the new mask compared to a traditional one (Visairo Mask).

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) is considered the gold standard treatment, in combination with medical therapy, for patients with respiratory acidosis secondary to Chronic Obstructive Pulmonary Disease (COPD). The choice of interface is a key factor in the success of NIV. A new oronasal mask, designed to improve CO2 washout (OptiNIV, Fisher & Paykel Healthcare, New Zealand), has recently been introduced to the market. Experimental data show that this interface, with a unique design separating airflow between the patient's mouth and nose, enhances gas flow at the end of expiration towards the oropharynx and subsequently out through the nostrils. This design facilitates the removal of CO2-rich air from the upper airways via dedicated ventilation ports located at the front of the mask, thereby optimizing CO2 clearance and dead space ventilation, which improves ventilatory efficiency.

This single-center, crossover study aims to investigate the effects of a new oronasal mask used during non-invasive ventilation (NIV) in COPD patients experiencing respiratory acidosis following an exacerbation. The objective is to assess whether the clinical benefits, specifically the reduction of PaCO₂ levels, are greater with the new mask compared to a traditional one. To minimize confounding factors affecting carbon dioxide washout, the new mask (OptiNIV, Fisher & Paykel Healthcare, New Zealand) will be compared to a mask of similar size, internal volume, and technical features (Visairo, Fisher & Paykel Healthcare, New Zealand), differing only in the presence of a separated airflow between the mouth and nose. This study holds significant clinical relevance, as no data are currently available on the use of the OptiNIV mask in patients with acute respiratory acidosis secondary to COPD exacerbation. The results could lead to optimized carbon dioxide clearance and improved ventilatory efficiency in managing patients with severe COPD exacerbations.

The study population consists of patients with respiratory acidosis secondary to COPD exacerbation who require non-invasive ventilation (NIV) and are admitted to the Respiratory and Critical Care Unit at the IRCCS AOU of Bologna, Policlinico S. Orsola. Patients meeting eligibility criteria will be randomly assigned (1:1) to two consecutive 60-minute NIV sessions using a traditional oronasal mask (Visairo) and an optimized mask (OptiNIV), following a crossover design. The sequence of mask use will be randomly assigned by the randomization list. NIV will be delivered with the same ventilator (ASTRAL 150 - ResMed Europe) using a single-limb circuit and pressure support mode, adjusting FiO₂ to maintain SpO₂ between 88-92%. Ventilator settings (IPAP, EPAP, triggers, rise time, Ti min, Ti max) will be set according to clinical practice but kept constant between sessions.

A 30-minute washout period with Venturi mask oxygen therapy will separate the two sessions, aiming to maintain SpO₂ between 88-92%. At the end of the washout, transcutaneous CO₂ (PtCO₂) will be measured; if this value is within ±2 mmHg of baseline, patient will proceed to the second session; otherwise, the washout will be extended up to 60 minutes. Including the washout, the total study duration per patient will not exceed 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed consent obtained
* Patients with COPD and acute hypoxemic-hypercapnic respiratory failure (pH < 7.35, PaO₂ < 60 mmHg, PaCO₂ > 45 mmHg) requiring non-invasive mechanical ventilation.

Exclusion Criteria:

* BMI ≥ 30 kg/m²
* Obstructive sleep apnea syndrome
* Neuromuscular diseases or chest wall pathologies
* Need for intubation and invasive mechanical ventilation during exacerbation
* Use of home non-invasive mechanical ventilation or CPAP
* Contraindications for NIV
* Cognitive disorders that may interfere with adherence to treatments
* Patients with active and unstable coronary artery disease
* Previous esophageal surgery, known esophageal stenosis, or any other condition that could put the patient at risk during the placement of the respiratory mechanics probe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effects of the OptiNIV oronasal mask on partial pressure of carbon dioxide (PaCO₂) levels in patients with severe COPD exacerbation requiring treatment with non-invasive mechanical ventilation. | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  Measured through arterial blood gas analysis. Unit of measurement: mmHg

SECONDARY OUTCOMES:
Evaluation of changes in paO2 | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured through arterial blood gas analysis Unit of measuremet: mmHg
Evaluation of changes in HCO3- | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured through arterial blood gas analysis
Evaluation of changes in pH | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured through arterial blood gas analysis
Evaluation of changes in PaO₂/FiO₂ | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured through arterial blood gas analysis
Evaluation of changes in blood pressure | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured using a sphygmomanometer Unit of measuremet: mmHg
Evaluation of changes in the heart rate | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured using a pulsoximeter Unit of measuremet: bpm
Evaluation of changes in the respiratory pattern | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured using the Minute Ventilation data and Respiratory Rate data obtained through a respiratory inductance plethysmography
Evaluation of changes in the Ventilatory Ratio | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured using the formula VR = (minute ventilation [ml/min] × PaCO₂) / (predicted weight [kg] × 100 × 37.5).
Evaluation of changes in the end-tidal carbon dioxide (etCO₂) | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured using a capnograph
Evaluation of changes in the esophageal pressure swing | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured via a nasogastric tube with an esophageal balloon.
Evaluation of changes in the asynchrony index | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured using the formula: AI = number of asynchronies / RR x 100 and will be measured by downloading the ventilator data at the end of each session
Evaluation of changes in transcutaneous SpO₂ % | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  Will be measured via transcutaneous monitoring of SpO₂ that will be performed using a dedicated device that will record data for the entire duration of the study. Data at the end of each session will be compared with the data obtained at the beginning of the session.
  Unit of measure: %
Evaluation of changes in transcutaneous TcCO2 | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  Will be measured via transcutaneous monitoring of TcCO2 that will be performed using a dedicated device that will record data for the entire duration of the study. Data at the end of each session will be compared with the data obtained at the beginning of the session.
  Unit of measure: mmHg
Evaluation of dyspnea | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured using a visual analog scale (VAS) ranging from 0 to 100 where 0 represents minimum dyspnea and 100 represents maximum dyspnea
Evaluation of the comfort level experienced | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  It will be measured using a visual analog scale (VAS) with a score ranging from 0 to 10, where 0 represents maximum comfort and 10 represents maximum discomfort.
Evaluation of NIV failure | T0 (baseline), T1 ( + 1 hour), T2 ( + 2 hours), T3 (+ 3 hours).
  NIV failure will be measured as the need for invasive mechanical ventilation (IMV)
Occurrance of adverse events | T1 ( + 1 hour) and at T3 (+ 3 hours).
  will be measured by recording any complications (skin irritation or ulcers, gastric distension, pneumothorax, hypotension, conjunctivitis, claustrophobia, aspiration) that occur during sessions with the two interfaces

CONTACTS AND LOCATIONS:
Locations (1):
- U.O Pneumologia e Terapia Intensiva Respiratora, IRCCS AOU di Bologna, Bologna, Bologna, Italy

REFERENCES:
- [Background] Piquilloud L, Olivier PY, Richard JC, Thepot-Seegers V, Brochard L, Mercat A, Beloncle F. High flow nasal cannula improves breathing efficiency and ventilatory ratio in COPD patients recovering from an exacerbation. J Crit Care. 2022 Jun;69:154023. doi: 10.1016/j.jcrc.2022.154023. Epub 2022 Mar 26. PMID 35349909
- [Background] Charususin N, Dacha S, Gosselink R, Decramer M, Von Leupoldt A, Reijnders T, Louvaris Z, Langer D. Respiratory muscle function and exercise limitation in patients with chronic obstructive pulmonary disease: a review. Expert Rev Respir Med. 2018 Jan;12(1):67-79. doi: 10.1080/17476348.2018.1398084. Epub 2017 Nov 6. PMID 29072087
- [Background] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265